CLINICAL TRIAL: NCT02139280
Title: A Prospective Randomized Trial Examining Low- or Intermediate-Dose Cyclophosphamide for Hematopoietic Stem Cell Mobilization in Patients With a Hematologic Malignancy
Brief Title: Cyclophosphamide for Hematopoietic Stem Cell Mobilization in Patients With a Hematologic Malignancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Kenneth Meehan, Director, Bone Marrow Transplant Program, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D13179
Record Dates: First submitted 2014-03-03; First posted 2014-05-15 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Hematologic Malignancies
Keywords: Cyclophosphamide; Hematopoietic; Stem Cell; Mobilization; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 2: Cyclophosphamide 3 gms/m(2) (Active Comparator): Patients will receive intravenous mesna 15 minutes prior to cyclophosphamide and again at 4 and 8 hours afterwards. Each infusion will be given over 15 minutes. Oral mesna can be substituted for the two post-cyclophosphamide doses. Oral mesna will be administered at 2 and 6 hours after the start of cyclophosphamide. Cyclophosphamide will be administered intravenously over one hour at the dose of 3 gms/m(2).
  Interventions: Drug: Cyclophosphamide
- Arm 1: 1.5 gms/m(2) Cyclophosphamide (Experimental): Patients will receive intravenous mesna 15 minutes prior to cyclophosphamide and again at 4 and 8 hours afterwards. Each infusion will be given over 15 minutes. Oral mesna can be substituted for the two post-cyclophosphamide doses. Oral mesna will be administered at 2 and 6 hours after the start of cyclophosphamide. Cyclophosphamide will be administered intravenously over one hour at the dose of 1.5 gms/m(2).
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Mechanism of action: Cyclophosphamide is a pro drug that requires activation. Following hepatic and cellular activation, phosphoramide mustard and acrolein are formed. Phosphoramide mustard is the alkylating agent that demonstrates cytotoxic effects. Acrolein binds to proteins but does not contribute to the anti-tumor effects.
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; Cytophosphane

SUMMARY:
No prospective randomized trials have evaluated the most efficacious dose of cyclophosphamide to mobilize autologous stem cells. We previously demonstrated that the time to collection of autologous hematopoietic stem cells is 10-12 days following the one dose of cyclophosphamide and daily G-CSF (granulocyte-colony stimulating factor).9 This prospective randomized trial is designed to determine if a lower dose of cyclophosphamide (1.5 gm/m2) will be as efficacious as the intermediate dose (3 gm/m2), based on cell number collected, number of apheresis required and resource utilization.

DETAILED DESCRIPTION:
This prospective randomized trial is designed to determine if a lower dose of cyclophosphamide (1.5 gm/m2) will be as efficacious as the intermediate dose (3 gm/m2), based on cell number collected, number of apheresis required and resource utilization.

The time to collection of autologous hematopoietic stem cells was ten to twelve days following cyclophosphamide and daily filgrastim. Peripheral blood CD34+ cell numbers were examined beginning ten days after cyclophosphamide administration. Leukapheresis began once the blood CD34+ number reached 10 cells/mcl. Patients received consecutive days of leukapheresis, with the goal of collecting > 5 x 106 CD34+cells/kg. The collection process, concentration and storage of PBSC were similar for all patients. Briefly, a 4-blood volume leukapheresis PBSC collection was performed daily using a COBE Spectra cell separator (COBE BCT, Lakewood, CO). Collected cells were concentrated and cryopreserved. Cells were frozen in Cryocyte freezing bags (Nexell Therapeutics Inc.) in a controlled rate freezer (Custom BioGenic Systems, Shelby Township, MI). At the conclusion of this freezing, the cells were transferred to the vapor phase of a monitored liquid nitrogen freezer (CryoPlus III, Forma Scientific, Marietta, OH) at a temperature of -120 0C or below.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a pathologic diagnosis of one of the following malignancies:

Non-Hodgkin's Lymphoma, including B- and T-cell lymphoma Multiple Myeloma or another plasma cell dyscrasia (Waldenstrom, Amyloidosis)

* The patient must be approved for transplant by the treating Transplant physician.
* This must be the patient's FIRST mobilization attempt.
* Patients are eligible if an autologous transplant is planned within approximately 12 months from the time of collection of cells.
* Prior Treatment: No previous cytotoxic chemotherapy within 4 weeks prior to initiation of therapy. (This does not include immunomodulatory drugs (IMiDs), proteasome inhibitors, monoclonal antibodies or steroids.)
* No radiation within 4 weeks of mobilization attempt.
* Age >18, and < 75 years
* No significant co-morbid medical or psychiatric illness that would significantly compromise the patient's clinical care and chances of survival.
* Informed consent must be signed prior to the treatment. Patients must willingly consent after being informed of the procedure to be followed, the nature of the therapy, alternatives, potential benefits, side effects, risks and discomforts. (Human protection committee approval of this protocol and a consent form is required.)

Exclusion Criteria:

* Medical, social, or psychological factors that would prevent the patient from receiving or cooperating with the full course of therapy.
* Documented hypersensitivity to any of the drugs used in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-12; Primary Completion 2019-07 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Meehan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 58 Individuals provided informed consent. Of those. four (4) participants were screen failures.
Period: Overall Study
Arm/Group | Arm 1: 1.5 Gms/m(2) Cyclophosphamide | Arm 2: Cyclophosphamide 3 Gms/m(2)
Started | 34 | 20
Completed | 32 | 20
Not Completed | 2 | 0
Not completed — No longer eligible | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: 1.5 Gms/m(2) Cyclophosphamide | Arm 2: Cyclophosphamide 3 Gms/m(2) | Total
Number analyzed (Participants) | 32 | 20 | 52
Age, Continuous [Median (Full Range); unit: years] | 62.5 [37 to 74] | 61.3 [51 to 74] | 61.9 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 21 | 10 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 32 | 20 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 20 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Nucleated Cells Collected Within the Apheresis Products
Description: the investigator will identify the number of cells collected within the apheresis products
Time Frame: 6 weeks
Measure: Median (Full Range); unit: cells x10e10
Arm/Group | Arm 1: 1.5 Gms/m(2) Cyclophosphamide | Arm 2: Cyclophosphamide 3 Gms/m(2)
Number analyzed (Participants) | 32 | 20
cells x10e10 | 5.7 [2.9 to 15.5] | 3.8 [1.9 to 7.1]

2. Primary Outcome: Number of CD34+ Cells Collected Within the Apheresis Products
Description: the investigator will identify the number of CD34+ cells collected within the apheresis products
Time Frame: 6 weeks
Measure: Median (Full Range); unit: cells x10e8
Arm/Group | Arm 1: 1.5 Gms/m(2) Cyclophosphamide | Arm 2: Cyclophosphamide 3 Gms/m(2)
Number analyzed (Participants) | 32 | 20
cells x10e8 | 7 [2.2 to 49.9] | 10.5 [1.9 to 29.4]

3. Secondary Outcome: Resource Utilization - Transfusions of Red Blood Cells
Description: Resources used during the mobilization and apheresis processes will be captured.
Time Frame: participants will be followed approximately 6 weeks following initiation of treatment
Population: Data was not collected due to the large geographic areas of the patient residence. It was too difficult to collect the date from multiple physicians from multiple states.
Arm/Group | Arm 1: 1.5 Gms/m(2) Cyclophosphamide | Arm 2: Cyclophosphamide 3 Gms/m(2)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Resource Utilization- Transfusion of Platelets
Description: Resources used during the mobilization and apheresis processes will be captured.
Time Frame: participants will be followed approximately 6 weeks following initiation of treatment
Population: as for outcome 3
Arm/Group | Arm 1: 1.5 Gms/m(2) Cyclophosphamide | Arm 2: Cyclophosphamide 3 Gms/m(2)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Resource Utilization- Hospitalizations
Description: Resources used during the mobilization and apheresis processes will be captured.
Time Frame: participants will be followed approximately 6 weeks following initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 1.5 Gms/m(2) Cyclophosphamide | Arm 2: Cyclophosphamide 3 Gms/m(2)
Number analyzed (Participants) | 32 | 20
Participants | 1 | 1

6. Secondary Outcome: Resource Utilization- Incidence of Febrile Neutropenia
Description: Resources used during the mobilization and apheresis processes will be captured.
Time Frame: participants will be followed approximately 6 weeks following initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 1.5 Gms/m(2) Cyclophosphamide | Arm 2: Cyclophosphamide 3 Gms/m(2)
Number analyzed (Participants) | 32 | 20
Participants | 2 | 2

7. Secondary Outcome: Toxicities During the Mobilization and Apheresis Processes
Description: Toxicities during the mobilization and apheresis processes Grade 3 and higher
Time Frame: participants will be followed approximately 6 weeks following initiation of treatment
Population: Number of participants who experienced a grade 3 or higher adverse event
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 1.5 Gms/m(2) Cyclophosphamide | Arm 2: Cyclophosphamide 3 Gms/m(2)
Number analyzed (Participants) | 32 | 20
Participants | 4 | 7

ADVERSE EVENTS:
Time Frame: Monitoring of toxicities will terminate on the last day of collection, since treatment-related toxicities occur during this time period. Patients who complete mobilization will be considered "off treatment" on the date of the last mobilization. There will be no specified follow up beyond the off treatment period other than following for engraftment. Average period of data collection was 10 days
Description: Evaluation of toxicities (other than Hematologic) will be graded using National Cancer Institute Common Toxicity Criteria, specifically CTC AE 4.0.
Arm/Group | Arm 1: 1.5 Gms/m(2) Cyclophosphamide | Arm 2: Cyclophosphamide 3 Gms/m(2)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/33 | 2/20
Other Adverse Events (participants affected / at risk) | 16/33 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: 1.5 Gms/m(2) Cyclophosphamide (N=33) | Arm 2: Cyclophosphamide 3 Gms/m(2) (N=20)
Infection (Infections and infestations) | 1 (1) | 2 (2) — Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: 1.5 Gms/m(2) Cyclophosphamide (N=33) | Arm 2: Cyclophosphamide 3 Gms/m(2) (N=20)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 5 (5) — BLOOD/BONE MARROW: Platelets
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pain: Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) — CARDIAC ARRHYTHMIA: Supraventricular and nodal arrhythmia - Sinus tachycardia
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — DERMATOLOGY/SKIN: Pruritus/itching: Vaginal pruritus
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain: Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain: Bone (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain NOS (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT02139280/Prot_SAP_000.pdf